CLINICAL TRIAL: NCT07095114
Title: A Phase I/II Study of Disappearing Markers for Daily Radiation Treatment Delivery
Brief Title: A Study of Disappearing Markers for Daily Radiation Treatment Delivery for Breast Cancer Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Michael Dominello, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-034
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Ductal Carcinoma in Situ; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magic Ink tattoo (Experimental): Magic Ink tattoo ink which is only visible when exposed to ultraviolet light will be used to mark radiation guidance
  Interventions: Other: Magic Ink

INTERVENTIONS:
Other: Magic Ink — A novel ink that is only visible when exposed to Ultraviolet light and can be hidden using white light will be inserted into the dermis to tattoo a radiation guidance tattoo into the skin of the participant

SUMMARY:
The goal of this clinical trial is to learn if tattoos applied with Magic Ink is as safe as commercially available standard tattoo ink for the purpose of radiation in women with breast cancer undergoing radiation treatment. The main questions are:

* Is the Magic Ink as safe as standard tattoo ink
* Does Magic Ink continue to function and remain visible for radiation therapists during the treatment Participants will be consented and given a skin assessment. Once enrolled participants will be administered the Magic Ink tattoo instead of the standard tattoo ink in preparation for their radiation treatment. Participants will also complete a survey regarding body image. Skin assessment will occur again after the first week of radiation and at 3 months later. Throughout the radiation therapy the medical physicist will complete surveys about ease of set-up of the equipment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed stage 0 ductal carcinoma in situ (DCIS), I, II or III breast cancer and be planning to undergo radiation therapy (RT) after surgery
* Participants must be 18 years of age or older
* Participant must be able to understand a written informed consent document and be willing to sign it
* Participant must be assigned female at birth
* Participant must have a Karnofsky performance score of greater than or equal to 70%
* Women of child bearing potential must agree to avoid becoming pregnant through defined periods during the course of RT and must meet one of the following:

  * Surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy
  * Post-menopausal, defined as no menses for at least 12 months prior to the screening visit without alternative medical causation
  * Agree to practice true abstinence from sexual intercourse
  * Not in a sexual relationship in which the may become pregnant (i.e., same-sex relationship)
  * If they are childbearing potential, agree to use at least one highly effective and at least one additional method of contraception.
* For the first six participants only: Participant must have a Fitzpatrick Skin Tone Scale of 5 or 6

Exclusion Criteria:

* Participants who have received prior radiation treatment to the affected breast.
* Participants with a history of allergic reaction or hypersensitivity attributed to any tattoo ink
* Participants with active chronic skin diseases such as psoriasis. Participants with inactive or controlled skin diseases are eligible for this study
* Participants that are pregnant or breastfeeding. If a participant wishes to participate in this study, breastfeeding should be discontinued
* Participants with a BMI greater than 44.5 as calculated within six months prior to the starting of the study. If there are multiple BMI measurements available in the chart, the most recent will be used to determine eligibility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
Safety of Magic Ink | 3 months after completion of Radiation Therapy
  Number of participants with treatment related adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0)

SECONDARY OUTCOMES:
Efficacy of Magic Ink | 3 months after the completion of Radiation Therapy
  Ease of radiation treatment (RT) setup. Participants will be categorized as "difficult" or "easy" setups. Difficult setups are setups with greater than 15% of the films for the treatment course result in a physician flag or reimaging based on clinically unacceptable or borderline acceptable setup.
Body Image Score | 3 months after the completion of Radiation Therapy
  Participants will complete a Body Image survey at baseline (prior to treatment) and 3 months after the completion of radiation therapy. The body image scale survey is a 10 question Likert scale where participants give a rating of Not at all, A little, Quite a bit or Very much. Responses will be compared to historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dominello, DO, Principal Investigator — Wayne State University
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No